CLINICAL TRIAL: NCT05730283
Title: Phase 2 Study of the Efficacy and Safety of ORC-13661 for the Prevention of Drug-Induced Hearing Loss in Patients Receiving Intravenous Amikacin Therapy for Pulmonary Non-Tuberculous Mycobacterium Disease
Brief Title: Prevention of Ototoxicity in NTM Patients Treated With IV Amikacin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Winthrop (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Oricula Therapeutics (Unknown); University of Washington (Other); National Jewish Health (Other); Mayo Clinic (Other); The University of Texas Health Science Center at Tyler (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor-Investigator, Kevin Winthrop, Professor, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SOUNDS Trial; U01DC020175 (NIH)
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Ototoxicity, Drug-Induced
Keywords: NTM; nontuberculous mycobacteria; ototoxicity; hearing loss
MeSH Terms: conditions — Ototoxicity; Hearing Loss | interventions — ORC-13661

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: If not specifically designated by protocol to be unblinded, all study patients, Sponsor, other entities and individuals will be blinded to study drug assignments. Site pharmacy personnel, one or more statisticians, patient dose monitor, and designated central project management personnel will be unblinded. Data Safety Monitoring Board (DSMB) members may choose to unblind themselves.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- High Dose ORC-13661 (Experimental): This arm is a daily treatment regimen of study drug (ORC-13661) with a loading dose of 150mg followed by a daily dose of 30mg. Treatment regimen will run concurrently with treatment with IV amikacin. Study drug treatment will continue until treatment with IV amikacin ends or 90 days, whichever is earlier.
  Interventions: Drug: ORC-13661
- Low Dose ORC-13661 (Experimental): This arm is a daily treatment regimen of study drug (ORC-13661) with a loading dose of 60mg capsules followed by a daily dose of 12mg capsules. Treatment regimen will run concurrently with treatment with IV amikacin. Study drug treatment will continue until treatment with IV amikacin ends or 90 days, whichever is earlier.
  Interventions: Drug: ORC-13661
- Placebo (Placebo Comparator): This arm is a daily treatment regimen of a placebo with a loading dose and a daily dose of placebo capsules to match the treatment arms. Placebo regimen will run concurrently with treatment with IV amikacin. Placebo regimen will continue until treatment with IV amikacin ends or 90 days, whichever is earlier.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORC-13661 — High-dose intervention (30mg daily)
  Arms: High Dose ORC-13661
Drug: ORC-13661 — Low-dose intervention (12mg daily)
  Arms: Low Dose ORC-13661
Drug: Placebo — Placebo intervention
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the effectiveness of the study drug, ORC-13361, in preventing hearing loss in patients with NTM infection who are undergoing treatment with IV amikacin therapy. The main question this study aims to answer is:

* Is ORC-13661 effective for preventing or lessening hearing loss induced by amikacin treatment?
* Is ORC-13661 effective for preventing or lessening other measures of hearing impairment?

Participants will be asked to take a study drug while they are being treated with IV amikacin. Participants will take study drug for 90 days or until the end of their amikacin treatment, whichever comes first. During this time, researchers will gather clinical data on the participants' health.

Researchers will compare three groups - two groups taking different doses of the study drug and one group taking a placebo drug - to see if dose of drug has any effect on preventing hearing loss. A placebo is a look-alike substance that contains no active drug.

DETAILED DESCRIPTION:
Nontuberculous mycobacteria (NTM) are environmental bacteria that can cause chronic, debilitating pulmonary disease, primarily affecting those over age 60. In more severe cases of NTM infection, patients are given a therapy with parenteral aminoglycoside antibiotics (AGs), to achieve control or cure. Amikacin is the most commonly used aminoglycoside for treatment in this setting, however it is limited by in its use by its tendency to cause ototoxicity including hearing loss and/or vestibular dysfunction. Ototoxicity refers to substances (i.e. medications) which are damaging to the inner ear sensory cells and may result in functional hearing loss and other negative effects.

This main goal of this study is to test the effectiveness of the study drug, ORC-13661, a small molecule compound being developed as an adjunct therapy to be administered during AG use in order to prevent associated ototoxicity. This study is a randomized, double-blind, placebo-controlled, multicenter, dose-ranging clinical trial to compare the effects and safety of ORC-13661 in preventing or mitigating hearing in patients taking amikacin.

105 participants will be enrolled across 5 enrolling sites over the course of the study. Participants will be randomized in equal numbers between three different study arms: high-dose ORC-13661, low-dose ORC-13661, and placebo. Participants will take study drug for 90 days from the start of their amikacin treatment or until their amikacin treatment ends, whichever comes first.

The primary outcome of this study is prevention or mitigation of amikacin-induced ototoxicity. Secondary outcomes include changes in speech perception, auditory and balance effects, and quality of hearing.

ELIGIBILITY:
Inclusion Criteria:

1. Providing informed consent, documented by signing and dating the currently valid informed consent form.
2. Considered by the Investigator to have unimpaired consent capacity, without reliance on a legally authorized representative.
3. Stated willingness and ability to comply with study procedures and availability for the duration of the study.
4. Aged > 18 and < 80.
5. NTM infection meeting current Pulmonary NTM guidelines from the American Thoracic Society and the Infectious Diseases Society of America (ATS/IDSA) for systemic (IV) aminoglycoside therapy.
6. Anticipated duration of IV amikacin treatment of at least 30 days at time of study entry.
7. Statement of ability to take oral medication and adhere to the daily dosing regimen.
8. For females of reproductive potential: If they are of childbearing potential, they must agree in writing to practice an effective double barrier method of contraception from the signing of the informed consent form until 1 month following discontinuation of study drug treatment or agree to practice true abstinence, when this is consistent with the preferred and usual lifestyle of the subject.
9. For males of reproductive potential: Agree to practice effective barrier contraception from the signing of the informed consent form until 3 months (one spermatogenesis cycle) following the last dose of study drug or agree to practice true abstinence.

Exclusion Criteria:

1. Received a systemic aminoglycoside antibiotic within 6 months prior to planned first dose of amikacin.
2. ECG at Screening or prior to randomization (mean of triplicate values) with QT interval corrected using Fridericia's formula (QTcF interval) ≥ 450 msec.
3. ECG at Screening or prior to randomization with abnormalities that, in the Investigator's judgment, might predispose patient to clinically significant arrhythmia.
4. Patients taking strong CYP3A4 inducers such as rifampin and rifabutin in the 7 days prior to randomization or have the need for ongoing treatment with concomitant oral or intravenous therapy with strong CYP3A4 inducers during the study. If an additional antibiotic is needed, then azithromycin will be used.
5. Patients taking strong CYP3A4 inhibitors such as clarithromycin in the 7 days prior to randomization or the need for ongoing treatment with concomitant oral or intravenous therapy with strong CYP3A4 inhibitors during the study. If an additional antibiotic is needed, then azithromycin will be used.
6. Patients taking clofazimine or bedaquiline AND who also have congestive heart failure, significant ventricular arrhythmia, uncorrected hypokalemia, or ECG (single at Screening, mean of triplicate prior to randomization) showing QRS > 120 msec or heart rate < 50 bpm.
7. Patients with amikacin exposure within the 6 months prior to randomization.
8. Patients with known amikacin resistance (MIC >64)
9. Progressive liver disease (Child-Pugh B or C) which would affect or invalidate interpretation of change from the baseline liver function tests over the course of the study.
10. Signs of disturbed integrity of the tympanic membrane, determined by otoscopy or tympanometry, including chronic perforation or middle ear or ear canal inflammation or effusion.
11. History of congenital hearing loss, otological surgery (excluding myringotomy tubes or simple tympanoplasty healed and currently intact), sudden hearing loss, or Meniere's disease.
12. Bilateral profound hearing loss (>90 Decibels [dB] HL) at all test frequencies.
13. Conductive hearing loss evidenced by average air-bone-gaps >15 dB HL for 0.25-4.0 kilohertz (kHz)
14. History of active malignancy, either untreated or under active treatment.
15. History of risk factors for Torsades des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
16. Venous access not adequate for performance of study procedures.
17. Presence of any circumstance, condition, ECG or laboratory finding that, based on investigator judgment, would interfere with study procedures or assessments or present to the patient an unreasonable risk from participation in this study.
18. Current or anticipated use of excluded concomitant medications as specified in Section 6.5.
19. Pregnant or lactating.
20. Female of childbearing potential who does not have a negative serum pregnancy test and does not agree in writing to using a double barrier method of contraception.
21. Female relying on menopausal status for contraception who does not have Follicle-Stimulating Hormone (FSH) level consistent with that condition and who does not agree in writing to using a double barrier method of contraception.
22. Currently under correctional supervision (imprisoned, on probation or parole).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Mitigation or Prevention of Ototoxicity | Baseline to 28 (±5) days after study treatment discontinuation or 28 days after 90 days of study treatment, whichever comes first.
  Outcome is measured by changes from baseline using the American Speech-Language-Hearing Association (ASHA) shift criterion in patients with NTM disease undergoing treatment with IV amikacin therapy

SECONDARY OUTCOMES:
Mitigation or Prevention of hearing impairment with regards to speech perceptions | Baseline to 28 (±5) days after study treatment discontinuation or 28 days after 90 days of study treatment, whichever comes first.
  Outcome is measured by changes to patient's speech perceptions using the High Frequency Digits-in-Noise (HF-DIN) test
Mitigation or Prevention of hearing impairment with regards to perceived auditory and balance effects | Baseline to 28 (±5) days after study treatment discontinuation or 28 days after 90 days of study treatment, whichever comes first.
  Outcome is measured by changes to patient's tinnitus using the Modified-Tinnitus Ototoxicity Monitoring Interview (TOMI)
Mitigation or Prevention of hearing impairment with regards to speech, spatial and quality of hearing | Baseline to 28 (±5) days after study treatment discontinuation or 28 days after 90 days of study treatment, whichever comes first.
  Outcome is measured by changes to patient's Speech, Spatial and Quality of Hearing Scale (SSQ12)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Winthrop, MD, MPH, Principal Investigator — Oregon Health and Science University; Edwin Rubel, PhD, Principal Investigator — Oricula Therapeutics
Locations (5):
- United States (5):
  - National Jewish Health, Denver, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chowdhury S, Owens KN, Herr RJ, Jiang Q, Chen X, Johnson G, Groppi VE, Raible DW, Rubel EW, Simon JA. Phenotypic Optimization of Urea-Thiophene Carboxamides To Yield Potent, Well Tolerated, and Orally Active Protective Agents against Aminoglycoside-Induced Hearing Loss. J Med Chem. 2018 Jan 11;61(1):84-97. doi: 10.1021/acs.jmedchem.7b00932. Epub 2017 Oct 27. PMID 28992413
- [Background] Garinis A, Gleser M, Johns A, Larsen E, Vachhani J. Prospective cohort study of ototoxicity in persons with cystic fibrosis following a single course of intravenous tobramycin. J Cyst Fibros. 2021 Mar;20(2):278-283. doi: 10.1016/j.jcf.2020.07.001. Epub 2020 Jul 24. PMID 32713806
- [Background] Gleser MA, Zettner EM. Negative hearing effects of a single course of IV aminoglycoside therapy in cystic fibrosis patients. Int J Audiol. 2018 Dec;57(12):917-924. doi: 10.1080/14992027.2018.1514537. Epub 2018 Nov 1. PMID 30382794
- [Background] Jarand J, Levin A, Zhang L, Huitt G, Mitchell JD, Daley CL. Clinical and microbiologic outcomes in patients receiving treatment for Mycobacterium abscessus pulmonary disease. Clin Infect Dis. 2011 Mar 1;52(5):565-71. doi: 10.1093/cid/ciq237. PMID 21292659
- [Background] Kitcher SR, Kirkwood NK, Camci ED, Wu P, Gibson RM, Redila VA, Simon JA, Rubel EW, Raible DW, Richardson GP, Kros CJ. ORC-13661 protects sensory hair cells from aminoglycoside and cisplatin ototoxicity. JCI Insight. 2019 Aug 8;4(15):e126764. doi: 10.1172/jci.insight.126764. eCollection 2019 Aug 8. PMID 31391343
- [Background] Potgieter JM, Swanepoel W, Smits C. Evaluating a smartphone digits-in-noise test as part of the audiometric test battery. S Afr J Commun Disord. 2018 May 21;65(1):e1-e6. doi: 10.4102/sajcd.v65i1.574. PMID 29781704
- [Background] Smits C, Theo Goverts S, Festen JM. The digits-in-noise test: assessing auditory speech recognition abilities in noise. J Acoust Soc Am. 2013 Mar;133(3):1693-706. doi: 10.1121/1.4789933. PMID 23464039
- [Background] Zettner EM, Gleser MA. Progressive Hearing Loss among Patients with Cystic Fibrosis and Parenteral Aminoglycoside Treatment. Otolaryngol Head Neck Surg. 2018 Nov;159(5):887-894. doi: 10.1177/0194599818782444. Epub 2018 Jun 19. PMID 29914288
- [Background] Carhart R, Jerger, J. Preferred method for clinical determination of pure-tone thresholds. J Speech Hear Disord. 1959; 24: 330-345.
- [Background] Kemp DT. Stimulated acoustic emissions from within the human auditory system. J Acoust Soc Am. 1978 Nov;64(5):1386-91. doi: 10.1121/1.382104. PMID 744838
- [Background] Chisholm J, Lacey C, Zalewski C, Christensen J, Wafa T, Kim J, Beri A, Fennelly K, Olivier K, Brewer C. Factors Influencing the Prevalence of Amikacin Ototoxicity. Poster presented at the National Center for Rehabilitative Research (NCRAR) Biennial Conference, Ototoxicity and Noise Damage: Translating Preclinical Findings to Audiological Management. 2019 September 25-27; Portland, Oregon.
- [Background] Lacey C, Chisholm J, Zalewski C, Christensen J, Wafa T, Kim HJ, Beri A, Olivier K, Fennelly K, Brewer C. Amikacin Ototoxicity: Risk Factors and Sensitivity of Grading Scales. Poster presented at The NIH Summer Poster Day. 2019 August 8; Bethesda, Maryland.
- [Background] Prasad K, Borre ED, Dillard LK, Ayer A, Der C, Bainbridge KE, McMahon CM, Tucci DL, Wilson BS, Schmidler GDS, Saunders J. Priorities for hearing loss prevention and estimates of global cause-specific burdens of hearing loss: a systematic rapid review. Lancet Glob Health. 2024 Feb;12(2):e217-e225. doi: 10.1016/S2214-109X(23)00514-4. PMID 38245112
- [Background] Bellairs JA, Redila VA, Wu P, Tong L, Webster A, Simon JA, Rubel EW, Raible DW. An in vivo Biomarker to Characterize Ototoxic Compounds and Novel Protective Therapeutics. Front Mol Neurosci. 2022 Jul 18;15:944846. doi: 10.3389/fnmol.2022.944846. eCollection 2022. PMID 35923755
- [Background] Owens KN, Santos F, Roberts B, Linbo T, Coffin AB, Knisely AJ, Simon JA, Rubel EW, Raible DW. Identification of genetic and chemical modulators of zebrafish mechanosensory hair cell death. PLoS Genet. 2008 Feb 29;4(2):e1000020. doi: 10.1371/journal.pgen.1000020. PMID 18454195